CLINICAL TRIAL: NCT01860248
Title: Topical Alkane Vapocoolant Spray Effectiveness On Arterial Puncture Pain Reduction In Emergency Department: Randomized Double Blind Placebo-Controlled Trial
Brief Title: Vapocoolant Spray Effectiveness On Arterial Puncture Pain: Randomized Double Blind Placebo-Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUMS 4341
Record Dates: First submitted 2013-05-07; First posted 2013-05-22 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Puncture Site Pain
Keywords: vapocoolant effectiveness; arterial puncture

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vapocoolant spray (Experimental): Vapocoolant is administered in 20 centimeters distance for 20 seconds to the patients as anesthetic before ABG.
  Interventions: Drug: Vapocoolant spray
- Water spray (Placebo Comparator): The Patients in this arm will receive water spray as anesthetic before ABG.
  Interventions: Drug: Water spray

INTERVENTIONS:
Drug: Vapocoolant spray — The Vapocoolant spray containing alkane is applied for 20 seconds.
  Other Names: Cryoanesthetic
  Arms: Vapocoolant spray
Drug: Water spray — This spray is covered so the patient and the investigator can not find the spray type out.
  Arms: Water spray

SUMMARY:
This study was aimed to compare pain levels from arterial blood gas (ABG) sampling performed with vapocoolant spray in comparison to placebo.

DETAILED DESCRIPTION:
Previous studies of vapocoolant sprays for reducing pain were mainly on venopuncture with inconsistent results. There was only one prospective open labeled controlled study on arterial blood gas sampling with ethyl chloride which did not show effectiveness. This study will assess the efficacy and tolerability of a topical alkane vapocoolant spray for arterial puncture in adults in comparison to control spray.

ELIGIBILITY:
Inclusion Criteria:

* age of 14 years or older,
* needs ABG as a part of their diagnosis

Exclusion Criteria:

* history of analgesic medication used within 24 hours of enrollment,
* any sign of decreased consciousness,
* history of skin hypersensitivity,
* inability to report a pain score,
* history of a known neurological problem that changes pain perception,
* history of cold related reactions (e.g. Raynaud's phenomenon, cold urticaria),
* abnormal Allen's test

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
puncture pain | 30 seconds after ABG
  30 seconds after ABG was performed, the patients would be asked about the puncture pain in verbal numerical pain scale.

SECONDARY OUTCOMES:
Vapocoolant application pain | 30 seconds affter procedure completion
  30 seconds after ABG was performed, the patients would be asked about the spray application pain in verbal numerical pain scale.
number of puncture attempts | 30 seconds after procedure
  The number of ABG sampling attempts is recorded 30 seconds after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shervin Farahmand, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini hospital complex, Tehran, Tehran Province, Iran